CLINICAL TRIAL: NCT03804801
Title: Effect of Hibiscus Sabdariffa on Blood Pressure in a University Population
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sulaiman AlRajhi Colleges (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SulimanAC-Hibiscus
Record Dates: First submitted 2019-01-07; First posted 2019-01-15 (Actual); Last update posted 2019-01-16 (Actual); Status verified 2019-01

CONDITIONS: Elevated Blood Pressure
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Intervention Model Description: The study participants will be randomized into 2 groups, one of which will receive the intervention and the other will not receive the intervention
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention Arm (or Group) (Experimental): This arm will receive the intervention (Hibiscus Sabdariffa extract supplement)
  Interventions: Dietary Supplement: Hibiscus Sabdariffa
- Control Arm (or Group) (No Intervention): This arm will receive no intervention whatsoever, not even placebo

INTERVENTIONS:
Dietary Supplement: Hibiscus Sabdariffa — The extract of the plant Hibiscus Sabdariffa, also known as sour or red tea
  Arms: Intervention Arm (or Group)

SUMMARY:
Hypertension, also known as high blood pressure, is a very common disease and is considered "the silent killer". Hypertension is responsible for at least 45% of deaths due to heart disease, and 51% of deaths due to stroke. Hypertension plays a part in the worry of heart disease, stroke and kidney failure and premature mortality and disability. If hypertension goes uncontrolled, in the long term, it will cause serious complications, most of which will necessitate costly interventions to be solved and managed. Apparently, these interventions may include cardiac bypass surgery, carotid artery surgery and dialysis, draining individual and government budgets. Recent studies show that hibiscus (Hibiscus sabdariffa) tea can lower blood pressure as effectively as some standard anti-hypertensive drugs can. Hibiscus is widely consumed around the world as a ruby-colored, lemony beverage. Hibiscus is safe and, unlike most blood pressure drugs, rarely causes side effects. All of the studies the investigators found in the literature were either underpowered or inconclusive. All of these studies recommended further studies with bigger samples to accurately assess the effect of hibiscus sabdariffa on blood pressure in hypertensive patients. The aim of this study is to assess the feasibility of a large-scale study assessing the effectiveness of Hibiscus sabdariffa on lowering blood pressure in individuals with elevated blood pressure.

DETAILED DESCRIPTION:
Research Question:

Will daily consumption of 240 ml of Hibiscus sabdariffa reduce blood pressure in individuals with elevated blood pressure?

Research Objectives:

Primary: To conduct a feasibility study investigating the effect of daily consumption of 240 ml of Hibiscus sabdariffa on blood pressure in individuals with elevated blood pressure

Secondary: To investigate the effect of daily consumption of 240 ml of Hibiscus sabdariffa on low-density lipoprotein (LDL) levels

Secondary: To investigate the effect of daily consumption of 240 ml of Hibiscus sabdariffa on sleep quality

Secondary: To investigate the effect of daily consumption of 240 ml of Hibiscus sabdariffa on stress levels

Trial Design:

This study is an open-label randomized controlled trial. The intervention arm is going to receive a 240 ml serving of hibiscus sabdariffa (sour tea) 1 time a day. The control arm will not have a placebo; hence, "open-label".

Allocation:

The investigators will use simple randomization in this trial. Each participant will have an assigned code number, which will be generated by a computer program, and then these numbers will randomly be placed into one of the two study arms by the same computer program. The participants will know to which study arm they belong to once the trial is officially started.

Study Setting:

This study will be conducted in Sulaiman Al-Rajhi Colleges (SRC) in Al-Qassim Region, Kingdom of Saudi Arabia

Interventions:

Participants will drink hibiscus sabdariffa 1 time a day for 3 months. Hibiscus sabdariffa will be given to the participants in the form of boxes filled with small paper bags filled with the herb (just like teabags). The participant will immerse the teabag in 240 milliliters of cold drinking water (the same volume as in a regular paper cup used for tea) and let it settle for 2-3 minutes before drinking it. This will be done 1 time a day for 3 whole months.

The participant will be given a month's supply on the first day of the trial, and additional supply will be given during the follow-up visits. Reminder text messages (SMS) will be sent regularly (every 2-3 days) to the participant to remind the participants of drinking the hibiscus. Regarding the study outcomes, the participant's blood pressure will be measured using a standardized manual sphygmomanometer at the times of measurement. Regarding the blood LDL levels, the participant will have a blood sample withdrawn and analyzed for LDL levels at the times of measurement. Regarding sleep quality and stress levels, the participant will fill out the respective questionnaires at the times of measurement.

Before initiating the trial, each participant will have the details of the trial, the benefits and risks of the intervention, and the possible outcome of the trial explained to the participants by one of the study investigators. To insure adherence to the intervention, participants in the intervention group will be sent either a text message (SMS) or an e-mail reminding the participants to take the hibiscus tea. The option of either SMS or e-mail depends upon the participant's preference. Any questions or concerns from the side of the participants will be cleared up before initiating the trial and during upcoming follow-up visits.

Multiple randomized controlled trials showed that ingestion of hibiscus tea significantly lowered blood pressure in hypertensive patients. Moreover, some studies showed that ingestion of hibiscus tea lowered LDL levels in addition to other positive changes in blood lipid profiles of patients. The investigators also want to assess if there is an effect of ingestion of hibiscus tea on sleep quality and stress levels.

Sample Size:

Sample size is based on feasibility trial, to test whether this can be done, not on sample size statistics. Also, the target population is pre-hypertensive individuals in a university setting (this includes students, teaching staff, administration staff, and workers). Since there is a definite effect of hibiscus on blood pressure, the investigators recognized that the investigators need a relatively small sample size for the investigators' trial. 40 subjects (randomized into two arms of 20 subjects each) is the required number of participants for the study in order to not comprise the statistical significance and power of the results.

Recruitment:

The principal investigators will invite subjects to participate in the study via sending e-mails to all university individuals. Individuals willing to participate in the trial will sign up to participate in the trial using an online registration form. The investigators used the definition of elevated blood pressure (pre-hypertension) given by the 2017 American Heart Association Guidelines: "Elevated blood pressure (pre-hypertension): Systolic blood pressure [SBP] between 120-129 mm Hg and diastolic blood pressure [DBP] less than 80 mm Hg." (15) The investigators also used the definition of essential hypertension given by the 2017 American Heart Association Guidelines: "Hypertension Stage I: Systolic blood pressure [SBP] 130 - 139 mm Hg OR diastolic blood pressure [DBP] 80 - 89 mm Hg. Hypertension Stage II: Systolic blood pressure [SBP] at least 140 mm Hg OR diastolic blood pressure [DBP] at least 90 mm Hg" (15) The target population is individuals with elevated or Stage I hypertensive levels of blood pressure. This means the investigators will be recruiting individuals with a systolic blood pressure of 120 - 139 mm Hg and a diastolic blood pressure of 80 - 89 mm Hg. After being recognized as eligible participants via the inclusion / exclusion criteria, these participants will be randomized into one of the two study arms.

Data Collection:

Blood pressure (the primary outcome) will be measured regularly during the trial; specifically, at the start of the trial, at 1 month after the official start, at 2 months after the official start, and at 3 months after the official start (at the end of the trial). Measurement will be done during curricular activity hours in the university clinic, on multiple days of each measurement week (to accommodate for the schedule differences of participants). The study investigators will measure each participant's blood pressure using a standardized sphygmomanometer.

Low-density lipoprotein [LDL] (a secondary outcome) will be measured twice during the trial; specifically, once at the official start of the trial, and once at 3 months after the official start (at the end of the trial). A blood sample will be drawn from the participant by the study investigators.

Sleep quality and stress levels (secondary outcomes) will be measured twice during the trial; specifically, once at the official start of the trial, and once at 3 months after the official start (at the end of the trial). The participant will fill out a validated questionnaire form regarding sleep quality (the Pittsburgh Sleep Quality Index [PSQI]) and another form regarding stress levels (the Depression, Anxiety, & Stress Scales [DASS] AND the Perceived Stress Scale [PSS]).

In addition, during each measurement point, the study investigators will inquire about the participants' adherence to the intervention and will ask about any possible adverse effects caused by the intervention. Time will be given to clear up any concerns or questions the participants may have regarding the trial or its details.

For follow-up, the participants will visit the study investigators at the official start of the trial, at 1 month after the official start, at 2 months after the official start, and at 3 months after the official start (at the end of the trial).

Statistical Methods:

The investigators will analyze the collected data using the IBM SPSS Statistics software. The investigators will use the latest version (Version 25).

The investigators will analyze the difference between the mean blood pressures of the intervention group prior to taking the hibiscus tea and the mean blood pressures of the intervention group after taking the hibiscus tea (at the end of the trial) using the paired t-tests. The investigators will analyze the difference between the mean blood pressures of the control group and the mean blood pressures of the intervention group (both before and after the intervention) using the unpaired t-tests.

Similarly, the difference between LDL levels of the control group and LDL levels of the intervention group will be analyzed via the unpaired t-tests.

The differences in sleep quality and stress levels between the control group and the intervention group will be analyzed using paired t-tests. The differences in sleep quality and stress levels in the intervention group before and after the intervention will be analyzed using paired t-tests as well.

Confidentiality:

Informed consent will be offered to every participant. The purpose of the study will be explained to all the participants and the investigators will ensure strict confidentiality and anonymity before proceeding with the study. The participants will be placed individually in the university clinic and only the investigators will record the results in order for the data collected to be totally confidential.

ELIGIBILITY:
Inclusion Criteria:

* Both sexes
* Age 18 - 70 years
* Abnormal blood pressure (SBP 120 - 139 mm Hg; DBP 80 - 89 mm Hg)
* Sulaiman Al Rajhi Colleges affiliate (student, teaching staff member, administrative staff member, worker)
* No regular medication

Exclusion Criteria:

* Allergic to hibiscus sabdariffa
* Normal blood pressure (SBP ≤ 120 mm Hg; DBP ≤ 80 mm Hg)
* Essential hypertension Stage II or higher (SBP ≥ 140 mm Hg; DBP ≥ 90 mm Hg)
* Hypertension due to secondary causes
* Other comorbid conditions (diabetes mellitus, renal failure, coronary artery disease, heart failure, malignant hypertension [BP ≥ 180/110], etc.)
* Regular hibiscus user
* Pregnancy
* Any metabolic or malabsorptive disease that may interfere with absorption of hibiscus sabdariffa (e.g. coeliac disease, chronic pancreatitis, etc.)
* Diagnosis of a sleep disorder or use of medication that interferes with sleep (either causing drowsiness or wakefulness)
* Diagnosis of a mood disorder or stress disorder
* Taking psychiatric medication (mood stabilizers, antidepressants, anxiolytics, or antipsychotics)

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2019-02-01 (Estimated); Primary Completion 2019-04-01 (Estimated); Study Completion 2019-06-29 (Estimated)

PRIMARY OUTCOMES:
Blood Pressure (BP) | 3 months
  The investigators want to see the effect of Hibiscus Sabdariffa on the blood pressure of participants in the intervention group.

SECONDARY OUTCOMES:
Low-density lipoprotein (LDL) levels | 3 months
  The investigators want to see the effect of Hibiscus Sabdariffa on the low-density lipoprotein (LDL) levels of participants in the intervention group.
The Pittsburgh Sleep Quality Index (PSQI) | 3 months
  The investigators want to see the effect of Hibiscus Sabdariffa on the sleep quality of participants in the intervention group.
  The Pittsburgh Sleep Quality Index (PSQI) contains 19 self-rated questions and 5 questions rated by the bed partner or roommate (if one is available). Only self-rated questions are included in the scoring. The 19 self-rated items are combined to form seven "component" scores, each of which has a range of 0-3 points. In all cases, a score of "0" indicates no difficulty, while a score of "3" indicates severe difficulty. The seven component scores are then added to yield one "global" score, with a range of 0-21 points, "0" indicating no difficulty and "21" indicating severe difficulties in all areas.
The Depression, Anxiety, and Stress Scales (DASS) | 3 months
  The investigators want to see the effect of Hibiscus Sabdariffa on the stress levels of participants in the intervention group.
  The DASS is a set of three self-report scales designed to measure the negative emotional states of depression, anxiety and stress.
  The DASS is composed of three 14-item subscales, for a total of 42 questions. DASS scores can be 0-42 on each subscale. Total score is calculated by summing the scores for each subscale.
  For each of the three subscales, a higher score indicates a more severe negative emotional state.
The Perceived Stress Scale (PSS) | 3 months
  The investigators want to see the effect of Hibiscus Sabdariffa on the stress levels of participants in the intervention group.
  Individual scores on the PSS can range from 0 to 40 with higher scores indicating higher perceived stress.
  * Scores ranging from 0-13 would be considered low stress.
  * Scores ranging from 14-26 would be considered moderate stress.
  * Scores ranging from 27-40 would be considered high perceived stress.

REFERENCES:
- [Background] Al-Shafei AI, El-Gendy OA. Effects of Roselle on arterial pulse pressure and left ventricular hypertrophy in hypertensive patients. Saudi Med J. 2013 Dec;34(12):1248-54. PMID 24343464
- [Background] Nwachukwu DC, Aneke EI, Obika LF, Nwachukwu NZ. Effects of aqueous extract of Hibiscus sabdariffa on the renin-angiotensin-aldosterone system of Nigerians with mild to moderate essential hypertension: A comparative study with lisinopril. Indian J Pharmacol. 2015 Sep-Oct;47(5):540-5. doi: 10.4103/0253-7613.165194. PMID 26600645
- [Background] Nwachukwu DC, Aneke E, Nwachukwu NZ, Obika LF, Nwagha UI, Eze AA. Effect of Hibiscus sabdariffaon blood pressure and electrolyte profile of mild to moderate hypertensive Nigerians: A comparative study with hydrochlorothiazide. Niger J Clin Pract. 2015 Nov-Dec;18(6):762-70. doi: 10.4103/1119-3077.163278. PMID 26289514
- [Background] Herrera-Arellano A, Miranda-Sanchez J, Avila-Castro P, Herrera-Alvarez S, Jimenez-Ferrer JE, Zamilpa A, Roman-Ramos R, Ponce-Monter H, Tortoriello J. Clinical effects produced by a standardized herbal medicinal product of Hibiscus sabdariffa on patients with hypertension. A randomized, double-blind, lisinopril-controlled clinical trial. Planta Med. 2007 Jan;73(1):6-12. doi: 10.1055/s-2006-957065. PMID 17315307
- [Background] Herrera-Arellano A, Flores-Romero S, Chavez-Soto MA, Tortoriello J. Effectiveness and tolerability of a standardized extract from Hibiscus sabdariffa in patients with mild to moderate hypertension: a controlled and randomized clinical trial. Phytomedicine. 2004 Jul;11(5):375-82. doi: 10.1016/j.phymed.2004.04.001. PMID 15330492
- [Background] Gurrola-Diaz CM, Garcia-Lopez PM, Sanchez-Enriquez S, Troyo-Sanroman R, Andrade-Gonzalez I, Gomez-Leyva JF. Effects of Hibiscus sabdariffa extract powder and preventive treatment (diet) on the lipid profiles of patients with metabolic syndrome (MeSy). Phytomedicine. 2010 Jun;17(7):500-5. doi: 10.1016/j.phymed.2009.10.014. Epub 2009 Dec 3. PMID 19962289
- [Background] Serban C, Sahebkar A, Ursoniu S, Andrica F, Banach M. Effect of sour tea (Hibiscus sabdariffa L.) on arterial hypertension: a systematic review and meta-analysis of randomized controlled trials. J Hypertens. 2015 Jun;33(6):1119-27. doi: 10.1097/HJH.0000000000000585. PMID 25875025
- [Background] Wahabi HA, Alansary LA, Al-Sabban AH, Glasziuo P. The effectiveness of Hibiscus sabdariffa in the treatment of hypertension: a systematic review. Phytomedicine. 2010 Feb;17(2):83-6. doi: 10.1016/j.phymed.2009.09.002. Epub 2009 Oct 3. PMID 19801187
- [Background] Buysse DJ, Reynolds CF 3rd, Monk TH, Berman SR, Kupfer DJ. The Pittsburgh Sleep Quality Index: a new instrument for psychiatric practice and research. Psychiatry Res. 1989 May;28(2):193-213. doi: 10.1016/0165-1781(89)90047-4. PMID 2748771
- See also: Ogden Publications, Inc., & Ogden Publications, Inc. (n.d.). Lower Blood Pressure Naturally With Hibiscus Tea — https://www.motherearthnews.com/natural-health/herbal-remedies/lower-blood-pressure-naturally-zmgz11zrog
- See also: Hibiscus: Uses, Side Effects, Interactions, Dosage, and Warning — https://www.webmd.com/vitamins/ai/ingredientmono-211/hibiscus
- See also: Hypertension Highlights 2017 - American Heart Association — https://www.heart.org/-/media/data-import/downloadables/hypertension-guideline-highlights-flyer-ucm_497841.pdf
- See also: Psychology Foundation of Australia - Overview of Depression, Anxiety, & Stress Scales (DASS) — http://www2.psy.unsw.edu.au/dass/over.htm
- See also: Depression, Anxiety, and Stress Scales (DASS) Questionnaire — http://www2.psy.unsw.edu.au/dass/Download%20files/Dass42.pdf